CLINICAL TRIAL: NCT06125288
Title: Assessment of Severity of Interstitial Lung Disease (ILD) in Children: Analytical Study of Risk Factors and Prognostic Parameters
Brief Title: Risk Factors and Prognostic Parameters of Interstitial Lung Disease in Children
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Reham kamal hamdi mohamed, assistant lecturer, Assiut University
Other Study IDs: ILD in children
Record Dates: First submitted 2023-11-06; First posted 2023-11-09 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Interstitial Lung Disease
MeSH Terms: conditions — Lung Diseases, Interstitial | interventions — Radiation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: lab investigation and radiation — 1. . Full history taking including
     * Environmental factors such as long term exposure to environmental hazards as bacteria, fungi, chemicals, tobacco smoke and air pollution.
     * Host factors Family history (you have a higher risk of ILD if a close relative has ILD). History of recurrent chest infection. History of exposure to medication such as radiation and chemotherapy. History of Multisystem autoimmune diseases
  2. Full examination general and systemic especially chest examination
  3. investigation
     * pulse oximetry.
     * lab investigation include complete blood count parameters .
     * radiological investigation including ( echocardiography - MSCT chest - chest -x ray

SUMMARY:
Study the severity and outcome of children with interstitial lung disease

DETAILED DESCRIPTION:
The child interstitial lung diseases (chILD) are a group of chronic lung diseases resulting from pathological changes of alveolar wall and capillary units.The epidemiology of the various forms of chILD is difficult to establish. small studies have suggested an approximate incidence of 0.5-0.8 cases per 100 000 children The prevalence is estimated to be 3.6 and 1.32 per million in the UK and Germany, respectively. but there are no recorded studies for its prevalence in Egypt due to the lack of standardized definitions , the inadequacy of organized reporting systems, and the variety of pathological conditions. In addition, clinical presentation is often nonspecific, contributing to a poor recognition of these disorders and confusion with other chronic pulmonary diseases .

childhood interstitial lung disease may be considered if the child meets at least three of the criteria presented (1) Respiratory symptoms (e.g., cough, difficult breathing, exercise intolerance). (2). Respiratory signs (e.g., retractions, tachypnea, clubbing, failure to thrive). (3). Hypoxemia. (4). Diffuse parenchymal abnormalities on chest imaging .

The causes of chILD often remain undetermined. These diffuse lung disorders are chronic, and often have high morbidity and mortality .

Mortality from childhood interstitial lung diseases ranges from 15 to 60% in different research reaching up to 100% in genetic and developmental causes.

There are many challenges and uncertainties for the early and correct diagnosis of interstitial lung disease in the pediatric patient. Three major challenges include, First , the fact that interstitial lung disease is less common in infants and children compared with adults. Therefore, most clinicians and radiologists are less familiar with considering and recognizing interstitial lung disease in this patient population.

Second, the clinical manifestations of interstitial lung disease particularly in infants and the young child are often subtle, highly variable, and typically nonspecific, such as dyspnea, tachypnea, crackles, and hypoxemia.

Lastly, there are currently no pathognomonic clinical or laboratory criteria for the diagnosis of interstitial lung disease in pediatric patients.

Some of the major uncertainties involving interstitial lung disease in this population include the decrease of information regarding the natural history of interstitial lung disease in childhood,the lack of understanding of the role of specific host factors in the pathogenesis of interstitial lung disease, and the absence of information on prognostic indicators in interstitial lung disease in childhood and more particularly in infants. Due to the above-stated challenges and uncertainties, evaluation and diagnosis of interstitial lung disease in childhood and particularly in infants has been markedly limited in the past.

Interstitial lung diseases may be classified a specific, suspicious, or non -specific diagnosis . A specific diagnosis was assigned to those cases in which a diagnosis was made with confidence based on careful consideration of clinical presentation , laboratory evaluations, and invasive diagnostic studies , such as lung biopsy.

A suspicious diagnosis was assigned to those cases in which the clinical presentation suggested a disorder (such as hypersensitivity pneumonitis from bird exposure) that could not be confirmed conclusively by diagnostic evaluation.

Non - specific diagnosis was assigned to those cases in which no specific or suspicious diagnosis could be made despite complete diagnostic evaluation.

The appropriate and definitive investigation are lung biopsy in order to establish a precise diagnosis so At our hospital, we face many obstacles regarding the diagnosis .

The present study will be on suspicious and specific groups

ELIGIBILITY:
Inclusion Criteria: All children more than 1 month and less than 18 years of age.

Suspected cases with:

1. tachypnea , Hypoxemia less than 90% in room air , rales and wheezes in absence of chest infection , retraction or deformed chest wall .
2. pulmonary hypertension by ECG or echocardiography.
3. x-ray and CT chest infiltrates.
4. Duration of illness more than 1 month.

Specific cases with:

1. symptoms and signs of suspected cases.
2. Lung biopsy.

   -

   Exclusion Criteria:• All children less than 1 month and more than 18 years
   * congenital heart disease.
   * bronchopulmonary dysplasia.
   * Telangiectasia.
   * Duration of illness less than 1 month

Ages: 1 Month to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: All children with suspected ILD that present to Assiut University Hospital Units
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
number of pediatric patient suffering from complication of interstitial lung disease at assiut university hospital. | baseline
  number of patiants present to assiut university with clinical complication (tachycardia -tachapnnea -dysnea - cyanosis ) and lab complication by complete blood count and radiological complication by ( chest x ray - chest msct -echocardiography).

CONTACTS AND LOCATIONS:
Overall Officials: Maher Mokhtar Ahmed, Professor, Study Director — asiut university hospital

REFERENCES:
- [Background] Fan LL, Kozinetz CA. Factors influencing survival in children with chronic interstitial lung disease. Am J Respir Crit Care Med. 1997 Sep;156(3 Pt 1):939-42. doi: 10.1164/ajrccm.156.3.9703051. PMID 9310017
- [Background] Clement A, Henrion-Caude A, Fauroux B. The pathogenesis of interstitial lung diseases in children. Paediatr Respir Rev. 2004 Jun;5(2):94-7. doi: 10.1016/j.prrv.2004.01.002. PMID 15135117
- [Background] Bush A, Cunningham S, de Blic J, Barbato A, Clement A, Epaud R, Hengst M, Kiper N, Nicholson AG, Wetzke M, Snijders D, Schwerk N, Griese M; chILD-EU Collaboration. European protocols for the diagnosis and initial treatment of interstitial lung disease in children. Thorax. 2015 Nov;70(11):1078-84. doi: 10.1136/thoraxjnl-2015-207349. Epub 2015 Jul 1. PMID 26135832